CLINICAL TRIAL: NCT07348965
Title: Pulsatile High-dose Furmonertinib in EGFR-mutant NSCLC With Leptomeningeal Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZF2025-387-01
Record Dates: First submitted 2025-12-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); Leptomeningeal Metastasis; Furmonertinib; EGFR Activating Mutation
Keywords: NSCLC; furmonertinib; leptomeningeal metastasis; cerebrospinal fluid
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): furmonertinib 320mg qod po
  Interventions: Drug: Furmonertinib 320mg qod po
- Cohort B (Other): furmonertinib 160mg qd po
  Interventions: Drug: Furmonertinib 160mg qd po

INTERVENTIONS:
Drug: Furmonertinib 320mg qod po — furmonertinib 320mg qod po until disease, progression or uncontrollable adverse reactions occur.
  Arms: Cohort A
Drug: Furmonertinib 160mg qd po — furmonertinib 160mg qd po until disease, progression or uncontrollable adverse reactions occur.
  Arms: Cohort B

SUMMARY:
The goal of this clinical trial is to clarify the efficacy and safety of the high-dose alternate-day furmonertinib in NSCLC with leptomeningeal metastasis. It will also explore the mechanism by which the high-dose alternate-day administration regimen enhances efficacy from a pharmacokinetic perspective, and investigate the impact of co-occurring mutations on the efficacy and prognosis of furmonertinib in the treatment of EGFR-mutant NSCLC with leptomeningeal metastasis. The main questions it aims to answer are:

Does the high-dose alternate-day administration regimen have definite efficacy? Does the high-dose alternate-day administration regimen have favorable safety? Does the high-dose alternate-day administration regimen improve efficacy by increasing the cerebrospinal fluid (CSF) concentration and CSF penetration rate of the drug? Which co-occurring mutations may affect the efficacy and prognosis of patients with EGFR-mutant NSCLC and leptomeningeal metastasis? Participants will enter Cohort A (320mg qod po) or Cohort B (160mg qd po) to receive furmonertinib based on their own willingness and the clinician's decision, until disease, progression or uncontrollable adverse reactions occur. All patients in Cohort A will undergo efficacy and safety evaluation, with some also participating in pharmacokinetic study; patients in Cohort B will only undergo pharmacokinetic study.

Efficacy and safety evaluation will be conducted through imaging examinations, neurological function assessment scales, quality of life self-assessment scales, and adverse event records. Pharmacokinetic study will be carried out by detecting the plasma concentrations and CSF concentrations of furmonertinib and its active metabolites, and calculating the CSF penetration rate for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-small cell lung cancer (NSCLC) confirmed by histopathological or cytopathological examination
2. Patients with EGFR exon 19 deletion or exon 21 L858R mutation
3. Patients with leptomeningeal metastasis (LMD) confirmed by positive cerebrospinal fluid (CSF) cytology (within 28 days prior to the first dose administration) and with at least 1 LMD lesion that can be repeatedly evaluated by magnetic resonance imaging (MRI)
4. Patients with disease progression after first-line tyrosine kinase inhibitor (TKI) treatment
5. Aged ≥18 years and ≤85 years, with no gender restrictions.
6. Sufficient organ function, defined as: absolute neutrophil count ≥ 1.5×10⁹/L, platelet count ≥ 75×10⁹/L, hemoglobin ≥ 90g/L total bilirubin ≤ 1.5×upper limit of normal (ULN) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (for patients with liver metastasis, total bilirubin can be relaxed to ≤ 3×ULN, and ALT/AST can be relaxed to ≤ 5×ULN) serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft-Gault formula)
7. For patients enrolled in the pharmacokinetic study: no prior treatment with furmonertinib (either in combination or as monotherapy)
8. Patients who have signed the informed consent form, are willing to receive treatment under this protocol, can adhere to medication administration, and have good compliance.

Exclusion Criteria:

1. Unable to complete the baseline assessment form
2. Complicated with severe or uncontrolled systemic diseases, including active infection, electrolyte disturbance, bleeding tendency, etc.
3. Pregnant or lactating women, or those with planned pregnancy during the study or within 6 months after the study ends
4. Presence of central nervous system complications requiring emergency neurosurgical intervention
5. Suffering from other malignant tumors or having a history of other malignant tumors
6. Complicated with severe brain diseases or mental illnesses that affect the patient's ability to report symptoms by themselves
7. Individuals without legal capacity, or those for whom medical or ethical reasons affect the continuation of the study
8. Other circumstances deemed unsuitable for participation in this study by the researcher.
9. Patients with a severe allergic diathesis, especially those who have experienced severe drug allergies or other serious adverse reactions during previous treatment with tyrosine kinase inhibitors (TKIs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
LM-DCR | From date of first administration of the study drug until the date of first documented leptomeningeal disease progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Leptomeningeal metastasis-disease control rate, calculated as the proportion of patients with leptomeningeal metastasis who achieve remission or stable disease, which will be determined based on the modified imaging assessment method formulated by the RANO-LM working group with imaging assessments.

SECONDARY OUTCOMES:
LM-ORR | From date of first administration of the study drug until the date of first documented leptomeningeal disease progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Leptomeningeal metastasis objective response rate, calculated as the proportion of patients with leptomeningeal metastasis who achieve remission, which will be determined based on the modified imaging assessment method formulated by the RANO-LM working group with imaging assessments.
neurological function | From date of first administration of the study drug until the date of first documented leptomeningeal disease progression or date of death from any cause, whichever came first, assessed up to 3 years.
  measured by NANO-LM standardized neurological examination
iDoR | From date of first administration of the study drug until the date of first documented leptomeningeal disease progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Intracranial duration of response means the time from the first achievement of intracranial disease remission to the first disease progression or death from any cause. Investigators will assess lesions other than leptomeningeal metastases according to the modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), while investigators and neuroradiological Independent Central Review (ICR) will evaluate the response of leptomeningeal metastases based on the modified neuroradiological criteria formulated by the RANO-LM working group.
iPFS | From date of enrollment until the date of first documented leptomeningeal disease progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Intracranial progression-free survival means the time from the date of enrollment to the first occurrence of intracranial disease progression or death from any cause. Investigators will assess lesions other than leptomeningeal metastases according to the modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), while investigators and neuroradiological Independent Central Review (ICR) will evaluate the response of leptomeningeal metastases based on the modified neuroradiological criteria formulated by the RANO-LM working group.
PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Progression-free survival means the time from the date of enrollment to the first occurrence of disease progression or death from any cause. Investigators will assess lesions other than leptomeningeal metastases according to the modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), while investigators and neuroradiological Independent Central Review (ICR) will evaluate the response of leptomeningeal metastases based on the modified neuroradiological criteria formulated by the RANO-LM working group.
OS | From date of enrollment until the date of death from any cause, assessed up to 5 years.
  Overall survival refers to the time from the date of enrollment to the date of death from any cause.
Quality of life evaluation | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Patient self-assessments of quality of life will be conducted using the Chinese versions of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 is a 30-item questionnaire comprising 5 functional scales, 3 symptom scales, 1 global health/QoL scale and 6 single items. The score of this questionnaire ranges between 1 and 4 in functional scales, symptom scales, and single items. The score ranges between 1 and 7 in global health/QoL scale. The higher score indicates the worse quality of life.
Quality of life evaluation | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Patient self-assessments of quality of life will be also conducted using the Chinese versions of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Brain Cancer Module (EORTC QLQ-BN20). The QLQ-BN20 is a 20-item questionnaire that assesses future uncertainty, visual disorder, motor dysfunction, and communication deficit, as well as seven single items (headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs, bladder control). The score of this questionnaire ranges between 1 and 4. The higher score indicates the worse quality of life.
AEs | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Adverse events will be recorded according to Common Terminology Criteria for Adverse Events version 6.0 (CTCAE v6.0)
CSF Penetration Rate | Patients will undergo twice of specimen collection: the first before treatment (-14 to 0 days) and the second 4 weeks after treatment (4weeks ±7 days).
  Cerebrospinal fluid penetration rate refers to the ratio of the drug's concentration in cerebrospinal fluid to its concentration in plasma.
Gene Mutation | at baseline and date of progression (assessed up to 3 years)
  Testing the gene mutation of plasma, CSF and the tumor tissue by NGS

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, M.D., Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol